CLINICAL TRIAL: NCT02172313
Title: Effect of Food on the Pharmacokinetics of Oral Semaglutide in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4154; 2013-004707-39 (EudraCT Number); U1111-1149-8127 (Other: WHO)
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fed conditions (Experimental): Fasting for 10 hours overnight followed by a high-fat, high-calorie meal, after the meal dosing of the tablet with 240 mL of water and a post-dose fasting period of 4 hours
  Interventions: Drug: semaglutide
- Fasting conditions (Experimental): Fasting for 10 hours overnight followed by dosing of the tablet with 240 mL of water and a post-dose fasting period of 4 hours
  Interventions: Drug: semaglutide
- Reference dosing condition (Experimental): Fasting for 6 hours overnight followed by dosing of the tablet with 120 mL of water and a post-dose fasting period of 30 min
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — For oral administration.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the effect of food on the pharmacokinetics (the exposure of the trial drug in the body) of oral semaglutide, in a SNAC (sodium N-[8-(2-hydroxybenzoyl) amino] caprylate) tablet formulation with three different dosing conditions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18-75 years (both inclusive) at the time of signing informed consent
* Body mass index of 18.5-29.9 kg/m^2 (both inclusive)
* A good general health based on medical history, physical examination, and results of vital signs, electrocardiogram and laboratory safety tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods. Female of child bearing potential must use effective methods of birth control for the duration of the trial and for 5 weeks following last dose of oral semaglutide. Only highly effective methods of birth control are accepted (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices)
* History of, or presence of, cancer, diabetes or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Not able or not willing to refrain from smoking or use of nicotine substitute products when staying at the clinical unit
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening
* Previous gastrointestinal surgery such as invasive and corrective procedures involving the oesophagus, stomach, duodenum, gallbladder, pancreas or intestinal resections. Exempt are subjects that underwent uncomplicated surgical and diagnostic procedures such as appendectomy, hernia surgery, polypectomy, biopsies, as wells as colonic- and gastric endoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration time curve | From time 0 to 24 hours after the 10th daily dose

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | 0 to 24 hours after the 10th daily dose
Time to maximum observed semaglutide plasma concentration | 0 to 24 hours after the 10th daily dose
Terminal half-life of semaglutide | After the 10th daily dose
Area under the SNAC (sodium N-[8-(2-hydroxybenzoyl) amino] caprylate) plasma concentration time curve | From time 0 to 24 hours after the 10th daily dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- [Derived] Baekdal TA, Breitschaft A, Donsmark M, Maarbjerg SJ, Sondergaard FL, Borregaard J. Effect of Various Dosing Conditions on the Pharmacokinetics of Oral Semaglutide, a Human Glucagon-Like Peptide-1 Analogue in a Tablet Formulation. Diabetes Ther. 2021 Jul;12(7):1915-1927. doi: 10.1007/s13300-021-01078-y. Epub 2021 Jun 2. PMID 34080123
- [Derived] Overgaard RV, Navarria A, Ingwersen SH, Baekdal TA, Kildemoes RJ. Clinical Pharmacokinetics of Oral Semaglutide: Analyses of Data from Clinical Pharmacology Trials. Clin Pharmacokinet. 2021 Oct;60(10):1335-1348. doi: 10.1007/s40262-021-01025-x. Epub 2021 May 10. PMID 33969456
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com